CLINICAL TRIAL: NCT06840067
Title: Single-arm Clinical Study of Carbon Ion Radiotherapy Combined with Nituzumab and Gemcitabine for Pancreatic Cancer.
Brief Title: Clinical Study of Carbon Ion Radiotherapy for Pancreatic Cancer.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gansu Wuwei Tumor Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 186698
Record Dates: First submitted 2025-02-10; First posted 2025-02-21 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-02

CONDITIONS: Pancreatic Cancer Metastatic; Pancreatic Cancer Non-resectable
Keywords: Carbon Ion Radiotheray; pancreatic cancer; Nimotuzumab; Gemcitabine
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Heavy Ion Radiotherapy; Drug Therapy

STUDY DESIGN:
Intervention Model Description: carbon ion radiotherapy (CIRT) combined with nituzumab and gemcitabine in the treatment of locally advanced and metastatic pancreatic cancer.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single-arm (Experimental): Study group
  Interventions: Radiation: carbon ion radiotherapy (CIRT)

INTERVENTIONS:
Radiation: carbon ion radiotherapy (CIRT) — 1.CIRT: GTV: Primary tumor visible on imaging and clinical examination, and involved regional lymph nodes identified by CT/MRI (≥1.0 cm) or PET/CT scan. CTV: GTV plus 5mm margin, include posterior peritoneal plexus area and elective node irradiation around the pancreas (ENI). PTV: CTV plus 2.5-5mm margin (depending on the system error of each unit; When pancreatic head cancer is close to the stomach and intestines, the gastrointestinal direction does not expand). ITV: delineated on 4D-CT considering the influence of respiratory activity. Prescription dose: Stratification by measuring the nearest distance between PTV and gastrointestinal tract (≥5mm or < 5mm); Pancreatic head cancer (distance < 5mm) : 52.8Gy(RBE)/4.4Gy/12Fx; Pancreatic head, body and tail cancer (≥5mm) : 57.2Gy(RBE)/4.4Gy/13Fx. CIRT was once a day, four or five times a week. 2.Chemotherapy:Gemcitabine 1000mg/m2, intravenous infusion, dl, d8; Q3w . 3.Targeted therapyNituzumab injection 400mg, Qw，at least 4-6 cycles.
  Other Names: targeted therapy; chemotherapy

SUMMARY:
The objective is to evaluate the efficacy and safety of carbon ion radiotherapy (CIRT) combined with nituzumab and gemcitabine in the treatment of locally advanced and metastatic pancreatic cancer.

DETAILED DESCRIPTION:
The objective is a single-center, single-arm, prospective Phase II clinical trial was conducted to evaluate the safety and efficacy of this regimen.

The primary criteria for inclusion were 18 to 80 years of age, histologically or cytologically confirmed pancreatic ductal adenocarcinoma, and clinician assessment as inoperable or patient rejection of manual surgery. All eligible patients will receive CIRT in combination with gemcitabine and nituzumab. The primary endpoint of the study was progression-free survival (PFS). All patients included in the study were followed for survival for at least 12 months. A safe and effective segmentation dose for pancreatic cancer suitable for our facility and RBE model was obtained. The comprehensive treatment of carbon ion radiation therapy, targeted therapy and chemotherapy is effective of refractory tumors, radiation-resistant tumors, and complex tumors. Using the physical dosimetry and biological advantages of heavy ions, we can improve the tumor control rate and reduce the occurrence of surrounding normal tissue damage, and provide new treatment suggestions for locally advanced and metastatic pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years and ≤80 years;
2. Indications: patients with locally advanced or metastatic pancreatic adenocarcinoma confirmed by histopathology or cytology (stage III - IV).
3. At least one measurable lesion was present according to RECIST version 1.1 evaluation criteria.
4. Suitable for one cycle of gemcitabine combined with nituzumab.
5. No history of other malignant tumors (except cured skin cancer and stage 0 cervical cancer);
6. Liver function, kidney function and bone marrow function were basically normal (ALT and AST < 1.5 times of high normal value (ULN), bilirubin < 1.5×ULN; Adult endogenous creatinine clearance rate of 60ml/min or serum creatinine SCR≤140μmoI/L, BUN≤6.8mmol/L; Hemoglobin level >9 g/dL; White blood cell count ≥3.0*109/L; Platelet count ≥100*109/L;)
7. Good physical condition, i.e. ECOG (Eastern United States Oncology Collaboration Group) 0~2; There were no complications such as severe pulmonary hypertension, cardiovascular disease, peripheral vascular disease, and severe chronic heart disease that may affect radiotherapy. Cardiac function grade 1. (According to the New York College of Cardiology Cardiac Function Scale (NYHA)
8. Adequate functions of major organs;
9. Predicted survival (after treatment) ≥3 months;
10. Informed consent has been signed by the patient or his legal representative before radiotherapy.

Exclusion Criteria:

1. Patients who have received monoclonal antibodies, EGFR-TKI therapy, anti-angiogenic drugs, and immunosuppressants within six months.
2. Patients with uncontrolled, cancerous pleural effusion requiring frequent drainage, pericardial effusion, or ascites (allowing for cytological confirmation of effusion), gastrointestinal bleeding, or those identified by the investigator as having a high blood risk within 14 days prior to admission.
3. Participated in other interventional clinical trials within 30 days prior to screening.
4. The dose limit for organs at risk cannot reach the preset safe dose limit.
5. Being on chronic steroid hormone therapy for more than 6 months (e.g., prednisone dose > 10 mg/ day or equivalent).
6. People who are allergic to the drugs or their ingredients used in this program.
7. Pregnancy (confirmed by serum or urine β-HCG test) or lactation
8. Persons with AIDS, including those who have received antiretroviral therapy; Active stage of syphilis;
9. Accompanied by serious comorbiditions, including uncontrolled systemic or co-existing diseases (pulmonary insufficiency, cardiovascular, pulmonary, liver, kidney, diabetes, etc.), drug or alcohol abuse, dependence, addiction, and/or mental illness that prevent the successful implementation of the trial protocol;
10. Patients with poor compliance, including those who may not be able to complete the treatment plan or receive prescribed follow-up and examination;
11. Patients had other malignant neoplasms (except cured skin cancer and stage 0 cervical cancer);
12. There are contraindications to radiotherapy;
13. having no or limited capacity for civil conduct;
14. Any medical history that, in the investigator's judgment, might interfere with the trial results or increase the patient's risk;
15. Any condition in which the physician considers that participation in the trial is not appropriate, the physician determines that the patient will not benefit from carbon ion radiotherapy, or that there are other co-existing conditions or other factors that may affect carbon ion therapy.
16. Inability to understand the purpose of treatment or unwillingness/inability to sign treatment consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
overall survival | 1 year
  overall survival（OS）

SECONDARY OUTCOMES:
Objective tumor response rate | 1 year
  Objective tumor response rate(ORR)
Progression-free survival | 1year
  Progression-free survival (PFS)

CONTACTS AND LOCATIONS:
Overall Officials: Xiaojun Li, Study Director — Gansu Wuwei Tumor Hospital
Locations (1):
- Heavy Ion Radiotherapy Department, Wuwei, Gansu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schultheis B, Reuter D, Ebert MP, Siveke J, Kerkhoff A, Berdel WE, Hofheinz R, Behringer DM, Schmidt WE, Goker E, De Dosso S, Kneba M, Yalcin S, Overkamp F, Schlegel F, Dommach M, Rohrberg R, Steinmetz T, Bulitta M, Strumberg D. Gemcitabine combined with the monoclonal antibody nimotuzumab is an active first-line regimen in KRAS wildtype patients with locally advanced or metastatic pancreatic cancer: a multicenter, randomized phase IIb study. Ann Oncol. 2017 Oct 1;28(10):2429-2435. doi: 10.1093/annonc/mdx343. PMID 28961832
- [Background] Arslan C, Yalcin S. Current and future systemic treatment options in metastatic pancreatic cancer. J Gastrointest Oncol. 2014 Aug;5(4):280-95. doi: 10.3978/j.issn.2078-6891.2014.030. PMID 25083302
- [Background] Hartimath SV, Alizadeh E, Solomon VR, Chekol R, Bernhard W, Hill W, Parada AC, Barreto K, Geyer CR, Fonge H. Preclinical Evaluation of 111In-Labeled PEGylated Maytansine Nimotuzumab Drug Conjugates in EGFR-Positive Cancer Models. J Nucl Med. 2019 Aug;60(8):1103-1110. doi: 10.2967/jnumed.118.220095. Epub 2019 Jan 17. PMID 30655327
- [Background] Shinoto M, Yamada S, Terashima K, Yasuda S, Shioyama Y, Honda H, Kamada T, Tsujii H, Saisho H; Working Group for Pancreas Cancer. Carbon Ion Radiation Therapy With Concurrent Gemcitabine for Patients With Locally Advanced Pancreatic Cancer. Int J Radiat Oncol Biol Phys. 2016 May 1;95(1):498-504. doi: 10.1016/j.ijrobp.2015.12.362. Epub 2015 Dec 20. PMID 26883565
- [Background] Shinoto M, Yamada S, Yasuda S, Imada H, Shioyama Y, Honda H, Kamada T, Tsujii H, Saisho H; Working Group for Pancreas Cancer. Phase 1 trial of preoperative, short-course carbon-ion radiotherapy for patients with resectable pancreatic cancer. Cancer. 2013 Jan 1;119(1):45-51. doi: 10.1002/cncr.27723. Epub 2012 Jun 28. PMID 22744973
- [Background] Hammel P, Huguet F, van Laethem JL, Goldstein D, Glimelius B, Artru P, Borbath I, Bouche O, Shannon J, Andre T, Mineur L, Chibaudel B, Bonnetain F, Louvet C; LAP07 Trial Group. Effect of Chemoradiotherapy vs Chemotherapy on Survival in Patients With Locally Advanced Pancreatic Cancer Controlled After 4 Months of Gemcitabine With or Without Erlotinib: The LAP07 Randomized Clinical Trial. JAMA. 2016 May 3;315(17):1844-53. doi: 10.1001/jama.2016.4324. PMID 27139057
- [Background] Loehrer PJ Sr, Feng Y, Cardenes H, Wagner L, Brell JM, Cella D, Flynn P, Ramanathan RK, Crane CH, Alberts SR, Benson AB 3rd. Gemcitabine alone versus gemcitabine plus radiotherapy in patients with locally advanced pancreatic cancer: an Eastern Cooperative Oncology Group trial. J Clin Oncol. 2011 Nov 1;29(31):4105-12. doi: 10.1200/JCO.2011.34.8904. Epub 2011 Oct 3. PMID 21969502
- [Background] Ciabatti S, Cammelli S, Frakulli R, Arcelli A, Macchia G, Deodato F, Cilla S, Giaccherini L, Buwenge M, Morganti AG. Radiotherapy of pancreatic cancer in older patients: A systematic review. J Geriatr Oncol. 2019 Jul;10(4):534-539. doi: 10.1016/j.jgo.2018.09.007. Epub 2018 Sep 28. PMID 30270196
- [Background] Kovac JD, Mayer P, Hackert T, Klauss M. The Time to and Type of Pancreatic Cancer Recurrence after Surgical Resection: Is Prediction Possible? Acad Radiol. 2019 Jun;26(6):775-781. doi: 10.1016/j.acra.2018.07.025. Epub 2018 Sep 22. PMID 30254003
- [Background] Riediger H, Keck T, Wellner U, zur Hausen A, Adam U, Hopt UT, Makowiec F. The lymph node ratio is the strongest prognostic factor after resection of pancreatic cancer. J Gastrointest Surg. 2009 Jul;13(7):1337-44. doi: 10.1007/s11605-009-0919-2. Epub 2009 May 6. PMID 19418101
- [Background] Siegel RL, Miller KD, Jemal A. Cancer statistics, 2020. CA Cancer J Clin. 2020 Jan;70(1):7-30. doi: 10.3322/caac.21590. Epub 2020 Jan 8. PMID 31912902